CLINICAL TRIAL: NCT01658813
Title: Phase II Trial of Chemoimmunotherapy With 5-Fluorouracil Followed by Interferon-alfa-2b in Previously-treated Metastatic Gastrointestinal, Kidney, or Lung Cancer
Brief Title: 5-Fluorouracil Followed by Interferon-alfa-2b in Previously-treated Metastatic Gastrointestinal, Kidney, or Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-09
Record Dates: First submitted 2012-08-02; First posted 2012-08-07 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-01

CONDITIONS: Gastrointestinal Cancer Metastatic; Renal Cell Cancer Metastatic; Non Small Cell Lung Cancer Metastatic
Keywords: Metastatic Gastrointestinal; Metastatic Kidney; Metastatic Lung
MeSH Terms: interventions — Fluorouracil; Interferons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5-Fluorouracil and Interferon (Experimental): 5-Fluorouracil
  Interferon-alfa-2b
  Interventions: Drug: 5-Fluorouracil and Interferon

INTERVENTIONS:
Drug: 5-Fluorouracil and Interferon — 5-Fluorouracil Interferon-alfa-2b
  Other Names: 5FU and Interferon

SUMMARY:
The purpose of this study is to determine whether the combination of a 5-Fluorouracil (5-FU) and interferon, which is able to stimulate the immune system to kill cancer cells, will help to increase tumor shrinkage in previously-treated metastatic gastrointestinal, kidney, or lung Cancer.

DETAILED DESCRIPTION:
Interferon with continuous infusion 5-Fluorouracil (5-FU) regimens have shown response rates ranging from 0-43% in various cancers. Monthly bolus 5-FU + interferon-alfa-2b has not undergone formal phase II testing. In a small pilot study, a 5 consecutive day schedule of 5-FU and interferon-alfa-2b resulted in the limiting toxicities of diarrhea and mucositis. A more limited schedule was recommended. Therefore, it is reasonable to examine such a schedule. In the current study, 5-FU will be followed by interferon-alfa-2b daily for 3 days to attempt to benefit from both the biochemical and immunologic mechanisms described above.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-proven, metastatic gastrointestinal, kidney, or lung cancer who have had disease progression on at least two prior systemic therapies.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 and estimated survival of at least 3 months.
* Patients must be felt to have recovered from effects of prior therapy, such as past expected white blood count nadir for chemotherapy (> 2 weeks for most agents, > 6 weeks for nitrosoureas or mitomycin-C)
* Patient consent must be obtained prior to entrance onto study.
* White blood count > 3500/mm3; platelet count of at least 100,000/mm3; hemoglobin > 9.0 gm/dl; bilirubin, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) less than 3 times the upper limit of normal; serum creatinine < 1.8.
* Corticosteroids and immunosuppressive agents are not permitted during the course of the study. Patients must have received no corticosteroids or immunosuppressive medications at least 2 weeks prior to entrance on-study.
* Patients with elevated temperatures > 100.5 degrees F, must have sources of occult infection excluded.
* Women of childbearing potential must have a negative pregnancy test and must take adequate precautions to prevent pregnancy during treatment.

Exclusion Criteria:

* Evidence of significant cardiovascular disease including history of recent (< 6 months) myocardial infarction, uncompensated congestive heart failure, primary cardiac arrhythmias (not due to electrolyte disorder or drug toxicity, for example) beyond occasional PVC's, angina, or cerebrovascular accident.
* Prior history of psychiatric disorder that could be exacerbated by interferon therapy or which could preclude completion of this therapy.
* Pregnancy or lactation.
* History of hypersensitivity to interferon alfa or fluoropyrimidines.
* History of severe debilitating pulmonary disease, such as chronic obstructive pulmonary disease requiring continuous oxygen therapy.
* History of autoimmune disease requiring immunosuppression.
* Documented inflammatory joint or systemic inflammatory disease (such as Lupus) which could be exacerbated by interferon therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Quan, MD, Principal Investigator — Western Regional Medical Center, Inc.
Locations (1):
- Western Regional Medical Center, Inc, Goodyear, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 5-FU and Interferon-alfa-2b: All patients received 5-Fluorouracil and Interferon-alfa-2b
Period: Overall Study
Arm/Group | 5-FU and Interferon-alfa-2b
Started | 18
Eligible | 18
Treated | 18
Completed | 15
Not Completed | 3
Not completed — Disease progression | 3

BASELINE CHARACTERISTICS:
Groups:
- Number of Participants: 5-Fluorouracil and Interferon-alfa-2b
Arm/Group | Number of Participants
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 57 [35 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS) was calculated as the time (months) from date of the start of treatment to the date of first observed disease progression (per standard Response Evaluation Criteria In Solid Tumors [RECIST] or date of death from any cause, whichever came first, assessed up to 2 years. The actual date of tumor assessments was used for this calculation. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of one or more new lesions.
Time Frame: Assessed up to 2 years
Population: Data was not collected
Groups:
- Progression Free Survival: 5-Fluorouracil and Interferon-alfa-2b
Arm/Group | Progression Free Survival
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Responses
Description: Radiographic studies to evaluate for response were done at 8 weeks (after 1 cycle). Standard RECIST response criteria were utilized. Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: up to 2 years.
Population: Data was not collected
Groups:
- Number of Responders: the number of patients responding
Arm/Group | Number of Responders
Number analyzed (Participants) | 0

3. Secondary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by radiographic imaging: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: up to 2 years
Population: Data was not collected
Groups:
- Response Rate: percentage of patients responding
Arm/Group | Response Rate
Number analyzed (Participants) | 0

4. Secondary Outcome: Median Duration of Response
Description: as for outcome 3
Time Frame: Up tp 2 years
Population: Data was not collected
Groups:
- Median Duration of Response: The median duration of response was determined.
Arm/Group | Median Duration of Response
Number analyzed (Participants) | 0

5. Secondary Outcome: Median Survival
Description: Median survival was measured from date of entry on study until date of death
Time Frame: up to 2 years
Population: Data was not collected
Groups:
- Median Survival: The median survival of patients treated on study was determined.
Arm/Group | Median Survival
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Number of Participants
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 18/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Number of Participants (N=18)
Rigors (General disorders) | 12
Nausea/emesis (Gastrointestinal disorders) | 10
Fever (General disorders) | 7
Fatigue (General disorders) | 6
Headache (General disorders) | 4
arthralgia/myalgia (General disorders) | 3
Catarrhal symptoms (General disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Aspartate aminotransferase elevation (Investigations) | 3
thrombocytopenia (Investigations) | 3
Leukopenia (Investigations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
anorexia (Metabolism and nutrition disorders) | 2
flu-like symptoms (General disorders) | 4
Anemia (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Gastroesophageal reflux (Gastrointestinal disorders) | 1
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
insomnia (Psychiatric disorders) | 1
Alanine aminotransferase elevation (Investigations) | 1
Alkaline phosphatase elevation (Investigations) | 1
malaise (General disorders) | 1
localized edema (General disorders) | 1
pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
sinus tachycardia (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No